CLINICAL TRIAL: NCT05069025
Title: Use of Music in Reducing Pain During Outpatient Hysteroscopy in Primarily Infertile Patients: Prospective Randomized Trial
Brief Title: Use of Music in Reducing Pain During Outpatient Hysteroscopy in Primarily Infertile Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Collaborators: Hospital El Gezeera (Other)
Responsible Party: Principal Investigator, Ahmed Samy aly ashour, assistant professor of obstetrics and gynecology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: a8233
Record Dates: First submitted 2021-09-25; First posted 2021-10-06 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Hysteroscopy
MeSH Terms: interventions — Music Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- music group (Experimental): In the music group, music chosen by the participant will be played through a speaker by the nursing staff during outpatient hysteroscopy. Music will be played through a speaker instead of headphones in order to maintain good communication and interaction between the participant and the doctor.
  Interventions: Other: music
- non-music group (Other): Participants in the non-music group will undergo outpatient hysteroscopy in the same setting and standard procedure without listening to any music.
  Interventions: Other: no-music

INTERVENTIONS:
Other: music — In the music group, music chosen by the participant will be played through a speaker by the nursing staff during outpatient hysteroscopy. Music will be played through a speaker instead of headphones in order to maintain good communication and interaction between the participant and the doctor.
  Arms: music group
Other: no-music — Participants in the non-music group will undergo outpatient hysteroscopy in the same setting and standard procedure without listening to any music.
  Arms: non-music group

SUMMARY:
The aim of this study is to demonstrate the value of music in outpatient hysteroscopy on patients' level of pain and satisfaction in primarily infertile patients.

ELIGIBILITY:
Inclusion Criteria:

* women with primary infertility requiring a diagnostic hysteroscopy as a part of an infertility diagnosis workup

Exclusion Criteria:

* women with suspected pregnancy

heavy vaginal bleeding recent pelvic infection those who received analgesics prior to OH a concomitant neurologic disease that could affect the correct evaluation of pain

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2021-10-10 (Estimated); Primary Completion 2022-04-10 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Intensity of pain | 5 minutes
  Pain intensity will be assessed by visual analogue scale during the procedure.visual analogue scale ranging from 0 to 10

SECONDARY OUTCOMES:
Intensity of pain | 30 minutes
  Pain intensity will be assessed by visual analogue scale 30 minutes after the procedure.visual analogue scale ranging from 0 to 10
women satisfaction | 30 minutes
  satisfaction will be assessed by visual analogue scale-like scale ranging from 0 to 10 (0=no satisfaction; 10=maximal satisfaction)

IPD SHARING:
Plan to Share IPD: Undecided